CLINICAL TRIAL: NCT01452997
Title: Evaluation of Topical Ibuprofen and Steroid in the Reduction of Local Reactions and Symptoms From an Aedes Aegypti Mosquito Bite
Brief Title: Evaluation of Anti-inflammatories in the Reduction of Bite Reactions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QA351
Record Dates: First submitted 2011-10-12; First posted 2011-10-17 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2013-03

CONDITIONS: Mosquito Bite
Keywords: mosquito; allergy; bite; ant-inflammatory; Aedes aegypti mosquito bite
MeSH Terms: conditions — Hypersensitivity; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibuprofen Gel (Active Comparator): Ibuprofen 5% gel
  Interventions: Drug: NSAI treatment
- Ibuprofen placebo (Placebo Comparator): K-Y jelly
  Interventions: Drug: NSAI treatment
- Eumovate (Active Comparator): 0.05% w/w clobetasone butyrate
  Interventions: Drug: Steroid treatment
- Cream Placebo (Placebo Comparator): Aqueous Cream B.P.
  Interventions: Drug: Steroid treatment

INTERVENTIONS:
Drug: NSAI treatment — Ibuprofen 5% gel
  Other Names: Fenbid gel
  Arms: Ibuprofen Gel; Ibuprofen placebo
Drug: Steroid treatment — Steroid intervention with 0.05% w/w clobetasone butyrate.
  Arms: Cream Placebo; Eumovate

SUMMARY:
The purpose of this study is to evaluate two separate antiinflammatory products for the relief of symptoms through suppression of the immunological and inflammatory response following a mosquito bite. The investigators have selected ibuprofen gel as a NSAI formulation and 0.05% Clobetasone butyrate as a steroid cream with their appropriate physical matched placebo products.

ELIGIBILITY:
Inclusion Criteria:

18 to 65 years of age (inclusive). Caucasian (white or pale skin) Good health as determined by medical history and physical examination Females of child bearing potential must confirm they are not pregnant at the study start and agree not to become pregnant throughout the duration of the study.

History of the following triad of symptoms following a previous mosquito bite: weal, flare, and pruritus as immediate reaction to mosquito bites at least once in the past (= mosquito bite sensitive stages III or IV).

Willingness to attend for all study procedures at designated intervals. Willingness to provide full consent to the study

Exclusion Criteria:

Abnormalities of the skin on the forearms (including sunburn) that might interfere with the study results, as determined by the investigator/clinician during physical inspection.

History of clinically significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, metabolic, or other disease deemed clinically significant by investigator / clinician Use of prohibited therapies (including cosmetics on either forearm) as specified in Section 6.3.3 of the Clinical Trial Protocol (use of systemic or local antihistamines, steroids, or NSAIDs during or within 2 weeks prior to planned date of first study procedure); use of any medication considered to have an influence on the outcome of the study.

Any acute illness within the 7 days prior to planned date of first study procedure which might interfere with the study results (as determined by the investigator/clinician from medical history).

History of malignancy within 5 years of the planned date of the first study procedure Neurological or psychiatric disease, or drug or alcohol abuse which would interfere with the subject's completion of the protocol assignments.

Participated in research involving an investigational drug within 3 months of the planned date of first study procedure.

History of known anaphylactic hypersensitivity to mosquitoes bites, bee or wasp stings.

History of allergic reaction to any of the topical agents used in the study or any of their components.

History of allergy to latex or other rubber material Women who are pregnant or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
size of wheal, flare in mm | 90 minutes
  The statistical difference between active and placebo agent on bite reaction measured as size of wheal, flare in mm and itching measured on a visual scale recorded by the subject.ct.

SECONDARY OUTCOMES:
Subjective pain and itching | 90 minutes
  Subjective record of pain and itching recorded on a visual scale

CONTACTS AND LOCATIONS:
Overall Officials: Ron Behrens, MD FRCP, Principal Investigator — London School of Hygiene and Tropical Medicine; James Logan, PhD, Study Director — London School of Hygiene and Tropical Medicine
Locations (1):
- London School of Hygiene and Tropical Medicine, London, United Kingdom